CLINICAL TRIAL: NCT01727206
Title: Open-label, Single-arm, Phase II, Prospective, Pilot Study of Tocilizumab in Patients With Erdheim-Chester Disease
Brief Title: Pilot Study of Tocilizumab in Patients With Erdheim-Chester Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Lorenzo Dagna, Professor, Ospedale San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECD-TCZ-01; 2012-003151-11 (EudraCT Number); GR-2009-1594586 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2012-11-12; First posted 2012-11-15 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Erdheim-Chester Disease
Keywords: Erdheim-Chester disease; Tocilizumab; Treatment; Phase II
MeSH Terms: conditions — Erdheim-Chester Disease | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tocilizumab (Experimental): Tocilizumab 8 mg/kg intravenously every month for six months
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab
  Other Names: Ro-Actemra; Actemra

SUMMARY:
The study we propose is a pilot phase II, interventional, treatment, open-label, single-arm, efficacy/safety clinical trial of a 6-month treatment with tocilizumab (8 mg/kg once monthly) in adult patients with extraskeletal Erdheim-Chester disease (ECD). Efficacy will be assessed as the effect of the treatment on the size of the measurable lesions, as evaluated by bidimensional measurements, and by the impact of the treatment on symptom control and on patient quality of life. Safety of the treatment will be determined by the analysis of adverse events and of the relevant safety laboratory parameters.

Secondary objectives of the study will be:

1. to better characterize the mechanisms underlying such disease and the possible response to the treatment. In particular: i) we will investigate the immunophenotypic and histomorphologic features of ECD histiocytes; ii) we will gather gene expression data from peripheral blood immune cells to better characterize their functional status, to define their transcriptional fingerprints and their possible modulation as a result of tocilizumab treatment; iii) we will assess the production of soluble mediators and the expression of activation molecules by monocytes derived from ECD patients, as well as after stimulation with selected inflammatory cytokines; iv) we will investigate the ex vivo and in vitro impact of tocilizumab treatment on those markers, for possible use as a predictor or indicator of response to treatment.
2. to investigate the metabolic pattern in ECD patients before and after tocilizumab treatment as evaluated by fluoro-d-glucose positron emission tomography (FDG-PET) and to verify if it can be an indicator of ECD activity.

ELIGIBILITY:
Inclusion Criteria:

* patients >= 18 years of age able to understand and sign an informed consent;
* histologically proven diagnosis of Erdheim-Chester disease ;
* an advanced disease not limited to the skeleton, with at least one measurable lesion;
* if females of childbearing potential, a negative pregnancy test and willingness to adhere to a highly effective contraceptive method of birth control for the duration of the study;

Exclusion Criteria:

* history of hypersensitivity to tocilizumab or to any of the excipients;

  ￼- severe infections requiring hospitalization or antibiotic therapy in the 30 days before the enrollment in the study;
* active tuberculosis, listeriosis, histoplasmosis, sepsis, abscesses, opportunistic infections; active hepatitis B or C virus infection;
* past history of tuberculosis (as documented by a positive purified protein derivative (PPD) skin test and/or a positive Quantiferon test and/or a chest X- ray), in the absence of a documented and appropriate administration of a specific treatment for latent tuberculosis;
* history of human immunodeficiency virus (HIV) infection;
* past history (< 5 years before enrollment) of a lymphoproliferative disorder or of a solid cancer (excluding cured basal cell or squamous cell carcinoma of the skin);
* moderate or severe heart failure (NYHA class III/IV), uncontrolled diabetes mellitus or other diseases that -according to the physician in charge of the protocol- may be of harm to the patient, if he/she would enroll in the study;
* history of alcohol and/or drug abuse;
* prior treatment with alkylating drugs (chlorambucil, cyclophosphamide);
* serum creatinine > 1.6 mg/dL in female patients or > 1.9 mg/dL in male patients, aspartate aminotransferase and/or alanine aminotransferase > 3 x upper limit of normal ; platelet < 100.000/fL; hemoglobin < 8.5 g/dL; white blood cell count < 1000/fL; lymphocyte < 500/fL; total bilirubin > 2.0 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-11; Primary Completion 2015-02 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Reduction in the dimensions of measurable lesions according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria | 6 months
Functional improvement in measurable indexes | 6 months
  Improvement in renal, hypophyseal, and respiratory function or of bone turnover, when altered at baseline
Variations of patient quality of life | 6 months
  As evaluated by standard questionnaires (HAQ, Short Form (SF)-36)
Analysis of the adverse events and of the relevant safety laboratory parameters | 6 months
  Monitoring of adverse events, variations in biochemical and hematological tests (full blood count, liver and renal function tests, lipid profile)
Variations in disease activity as evaluated by FDG-PET imaging | 0, 2 and 6 months

SECONDARY OUTCOMES:
Evaluation of soluble factors, receptors and activation molecules involved the accumulation, activation and entrapment of histiocytes possibly associated to a response to the experimental treatment | 6 months
  * the levels of circulating cytokines and chemokines before, during and after tocilizumab treatment;
  * the immunophenotype and the transcriptional fingerprints of circulating immune cells from ECD patients and their possible modulation as a result of tocilizumab treatment;
  * the pathways involved in the production of interleukin (IL)-6 and IL-6-induced cytokines and chemokines by mononuclear cells obtained from ECD patients;
  * the interference of tocilizumab in vitro on monocyte activation and ex vivo from treated patients, also to evaluate its effect on the profile of circulating cytokines and on the secretory potential of patient-derived monocytes

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Dagna, MD, Principal Investigator — San Raffaele Scientific Institute
Locations (1):
- San Raffaele Hospital, Milan, Italy